CLINICAL TRIAL: NCT06898099
Title: Evaluation of the Efficacy of E2R Hypnotherapy in the Management of Chronic Insomnia in Primary Care
Brief Title: Evaluation of the Efficacy of E2R Hypnotherapy in the Management of Chronic Insomnia in Primary Care (HypERR)
Acronym: HypERR
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rennes University Hospital (Other)
Collaborators: Rennes University (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 35RC22_8973_HypERR; 2024-A01366-41 (Registry Identifier: ID-RCB_ANSM)
Record Dates: First submitted 2025-03-20; First posted 2025-03-27 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Chronic Insomnia
Keywords: chronic insomnia; E2R hypnosis; emotion-focused therapy; primary care; general medicine
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: The HypERR study is a multicenter, randomized, open-label study designed to confirm the efficacy of a hypotherapy method called E2R in the management of chronic insomnia, by comparing it with standard care (without hypnosis)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard care (Active Comparator): Patients will receive the usual care offered by their GP, the investigator in the study (except hypnosis).
  Interventions: Other: "Standard care" control group (without hypnosis)
- E2R hypnosis (Experimental): 4 x 30-minute hypnotherapy sessions over 6 weeks by the hypnotherapist using the E2R method (with self-hypnosis)
  Interventions: Other: Experimental group: "E2R hypnosis"

INTERVENTIONS:
Other: "Standard care" control group (without hypnosis) — Randomization stratification on insomnia severity. In the "Standard care" group, the investigating physician will not change his or her current practice as part of the study. Treatment will be the same as usual, whether drug-based or not (psychotherapy, etc.), with the exception of hypnosis. The patients will be reviewed at 3 months and 6 months (+/- 1 week) after randomization (D0). The following study information and questionnaires will be completed according to patients' responses: ISI and PSQI self-questionnaires, Record of psychotropic medications, Record of any non-drug therapies implemented, Events that could modify sleep, Serious adverse events (EvIG) and non-serious adverse events (EvING) of a neuropsychiatric nature that occurred or worsened during the study.
  Arms: Standard care
Other: Experimental group: "E2R hypnosis" — Randomization stratification on insomnia severity. For the patients randomized to the Hypnosis E2R arm, patients summoned within 15 days to 3 weeks of inclusion for their first hypnotherapy session with the hypnotherapist. All patients will receive 4 hypnotherapy sessions over 6 weeks using the E2R method.
  The patients will be reviewed at 3 months and 6 months (+/- 1 week) after randomization (D0). The following study information and questionnaires will be completed according to patients' responses: ISI and PSQI self-questionnaires, Record of psychotropic medications, Record of any non-drug therapies implemented, Practice of self-hypnosis requested of the patient (patient diary), Events that could modify sleep, Serious adverse events (EvIG) and non-serious adverse events (EvING) of a neuropsychiatric nature that occurred or worsened during the study.
  Arms: E2R hypnosis

SUMMARY:
In France, the treatment of chronic insomnia relies mainly on hypnotic drugs in routine care, despite the high level of iatrogenicity. Cognitive-behavioral therapy (CBT) is recommended by the HAS as a non-pharmaceutical first-line therapy for chronic insomnia. Despite evidence of their efficacy in chronic insomnia, these therapies remain underdeveloped in France (few practitioners, time-consuming for the patient). Hypnotherapy is another non-drug intervention suitable for routine outpatient care. Among the hypnosis methods practiced in France, E2R (Emotion, Regression, Repair) is a hypnotherapy method used in general practice, particularly for chronic insomnia. To date, no clinical trials have been carried out to demonstrate its effectiveness in this pathology.

The HypERR study is a multicenter, randomized, open-label study designed to evaluate the efficacy of a hypotherapy method called E2R in the management of chronic insomnia, by comparing it with standard care (without hypnosis).

DETAILED DESCRIPTION:
The selection and inclusion of patients will be carried out by 34 GPs (General Practitioner), the study investigators. They will then randomize their patients into one of 2 groups: the E2R hypnosis group versus the "standard care" control group (without hypnosis).

Patients randomized to the hypnosis group will be referred by their GP to a hypnotherapist in their area within a 30-minute radius. They will receive 4 x 30-minute hypnotherapy sessions over 6 weeks.

For patients randomized to the control group, the GP will be free to implement psychotherapy and/or other non-medication interventions as usual (with the exception of hypnosis) and/or medication.

Then, all patients will be reviewed at 3 and 6 months by their GP (+/- 1 week) after randomization (D0) to assess the study criteria.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 18 or over,
* Patient suffering from chronic insomnia according to the DSM-5 definition, whether or not treated with psychotropic drugs:

  * At least one of the following sleep disorders: difficulty in falling asleep, difficulty in maintaining sleep, waking up too early and inability to go back to sleep, and * At least 3 nights a week for at least 3 months, and * In an adequate night-time sleep context, and * With at least one significant impact on, or impairment of, social, occupational or behavioral functioning, and * Insomnia not attributable to the physiological effects of a substance, and * Insomnia not explicable by a medical condition or mental disorder.
* Patient willing to undergo hypnotherapy for 4 sessions of 30 min over 6 weeks,
* Patient whose treating physician is the investigator,
* Patient able to give free, informed, written consent,
* Patient affiliated to the French social security system.

Exclusion Criteria:

* Patients receiving or having received one or more hypnotherapy sessions (for any reason) in the last 5 years prior to inclusion,
* Patient participating in another study involving the treatment of insomnia or another pathology having an impact on sleep disorders,
* Patient unable to complete a self-administered questionnaire,
* Patients with poor or no understanding of the French language,
* Patients unable to attend hypnotherapy consultations,
* Deaf or hard-of-hearing patients without hearing aids,
* Patient under legal protection (safeguard of justice, curatorship, guardianship) or deprived of liberty,
* Women declaring themselves pregnant or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Estimated)
Dates: Start 2025-09-15 (Estimated); Primary Completion 2027-03-15 (Estimated); Study Completion 2027-03-15 (Estimated)

PRIMARY OUTCOMES:
Severity of Insomnia assessed by the Insomnia Severity Index (ISI) | 6 months
  Insomnia Severity Index (ISI). The minimum score is 0 meaning No Insomnia, the maximum is 28 meaning Severe clinical insomnia

SECONDARY OUTCOMES:
Severity of Insomnia assessed by the Insomnia Severity Index (ISI) | 3 months
  Insomnia Severity Index (ISI). The minimum score is 0 meaning No Insomnia, the maximum is 28 meaning Severe clinical insomnia
Number of responders assessed by the Insomnia Severity index (ISI) | 3 months
  The responders are defined by a decrease > 7 points on the ISI scale
Number of responders assessed by the Insomnia Severity index (ISI) | 6 months
  The responders are defined by a decrease > 7 points on the ISI scale
Number of partial responders assessed by the Insomnia Severity index (ISI) | 3 months
  Partial responders are defined by a decrease between 4 and 7 points on the ISI scale)
Number of partial responders assessed by the Insomnia Severity index (ISI) | 6 months
  Partial responders are defined by a decrease between 4 and 7 points on the ISI scale)
Number of non-responders assessed by the Insomnia Severity index (ISI) | 3 months
  Non-responders are defined by a decrease < 4 points on ISI scale
Number of non-responders assessed by the Insomnia Severity index (ISI) | 6 months
  Non-responders are defined by a decrease < 4 points on ISI scale
Consumption of Benzodiazepine and related drug assessed by the prescription and patient interview | 3 months
  Benzodiazepine and related drug consumption recorded by the investigator (prescription and patient interview).
Consumption of Benzodiazepine and related drug assessed by the prescription and patient interview | 6 months
  Benzodiazepine and related drug consumption recorded by the investigator (prescription and patient interview).
Sleep quality assessed by the Pittsburg Sleep Quality Index (PSQI) | 3 months
  Pittsburg Sleep Quality Index (PSQI self-questionnaire). The minimum score is 0 meaning no difficulty, the maximum score is 21 indicating major difficulties
Sleep quality assessed by the Pittsburg Sleep Quality Index (PSQI) | 6 months
  Pittsburg Sleep Quality Index (PSQI self-questionnaire). The minimum score is 0 meaning no difficulty, the maximum score is 21 indicating major difficulties
Incidence of neuropsychiatric Non-Serious Adverse Events (Safety) of E2R hypnosis method in primary care | 6 months
  Number and nature of neuropsychiatric Non-Serious Adverse Events (NSEs) that occurred or worsened during the study period.
Incidence of Serious Adverse Events (Safety) of E2R hypnosis method in primary care | 6 months
  Number and nature of Serious Adverse Events (EvIG) over the follow-up period

CONTACTS AND LOCATIONS:
Overall Officials: Eric MENER, Ph D, Principal Investigator — University of Rennes (Department of general practice)
Locations (30):
- France (30):
  - Cabinet médical, Bain-de-Bretagne
  - Cabinet médical de Plaisance, Bouaye
  - Cabinet médical de Breteil, Breteil
  - Cabinet médical, Cesson-Sévigné
  - Cabinet médical du Linon, Combourg
  - Cabinet médical Sycamore, Contres
  - Cabinet médical de Corps Nuds, Corps-Nuds
  - Cabinet médical des Embruns, Crac'h
  - Pôle Santé Physiomast, Dol-de-Bretagne
  - Maison médicale, Iffendic
  - Cabinet Médical Chantepie, Joué Les Tours
  - Cabinet Médical de Jugon-Les-Lacs -Saint-Igneuc, Jugon-les-Lacs
  - Maison médicale des Longrais, La Chapelle-des-Fougeretz
  - Cabinet médical, La Chapelle-Saint-Ursin
  - Cabinet médical du Lion d'Or, Nantes
  - Maison médicale Laennec, Pleudihen-sur-Rance
  - Maison De Santé De Ronsouze, Ploërmel
  - Cabinet médical Les Petits Ponts, Pont-Saint-Martin
  - Maison de Santé de Questembert, Questembert
  - Cabinet médical Olec, Rennes
  - Cabinet médical, Rennes
  - Maison médical de Maen roch, Saint-Brice-en-Coglès
  - Maison médicale, Saint-Gilles-Croix-de-Vie
  - Maison de soin du Couesnon, Saint-Ouen-des-Alleux
  - Cabinet médical, Saint-Romain-sur-Cher
  - Maison de santé, Sancerre
  - Cabinet médical de la Blanchisserie, Sully-sur-Loire
  - Maison de santé, Talensac
  - Cabinet des médecins généralistes de TIGY, Tigy
  - Cabinet médical, Vildé-Guingalan

IPD SHARING:
Plan to Share IPD: Yes
After informing patients, In accordance : data protection provisions (GDPR and French Data Protection Act) :
  Intention to share individual data All individual data collected during the study, after pseudonymization and minimization Protocol, amendments, observation log, information sheet and research consent form, statistical analysis plan, statistical analysis code, statistical report, study report without personal data, list of tables, variables and their definitions Data availability : Immediately after publication of the main analysis results and until the database is deleted Data recipients: Project leaders whose reuse has been approved by the sponsor (owner of the study data) and by the study steering committee Types of analyses: Analyses enabling the objectives defined in the sharing agreement to be achieved, which will be drawn up at the time of sharing Access via data request form sent to the promoter and data sharing agreement signed before any data is made available